CLINICAL TRIAL: NCT07301463
Title: A Multicenter, Longitudinal, Observational Study in Children With Achondroplasia
Brief Title: A Study in Children With Achondroplasia
Status: Recruiting | Type: Observational
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ABSK061-001
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Achondroplasia: Male or female aged ≥2.5 to <11 years old at screening
  Interventions: Other: No Interventions; Other: complete a natural history observation of ACH for at least 6 months and up to 2 years

INTERVENTIONS:
Other: No Interventions — No Interventions
Other: complete a natural history observation of ACH for at least 6 months and up to 2 years — no interventions

SUMMARY:
The goal of this observational study is to collect the anthropometric parameters, clinical characteristics, related medical complications, health-related quality of life and treatments of children with ACH, and complete a natural history observation of ACH for at least 6 months and up to 2 years.

DETAILED DESCRIPTION:
Primary Objectives To evaluate the safety, tolerability, and recommended dose for expansion (RDE) of oral ABSK061 in children with ACH To evaluate the efficacy of oral ABSK061 in children with ACH

Secondary Objectives To characterize the pharmacokinetics (PK) of ABSK061 and potential disproportional metabolites (if applicable) To evaluate changes from baseline in anthropometric parameters after administration of oral ABSK061 To evaluate the acceptability of ABSK061 minitablets for peroral administration in children with ACH

Exploratory Objectives To evaluate changes in ACH complications and disease burden after oral administration of ABSK061 To evaluate the pharmacodynamic (PD) profile in children with ACH after oral administration of ABSK061

ELIGIBILITY:
Inclusion Criteria:

1. Prior to screening, the guardians and children with ACH (if applicable) must be willing and able to provide signed informed consent.
2. Clinical diagnosis of ACH confirmed FGFR3 mutation by genetic testing.
3. Male or female aged ≥2.5 to <11 years old at screening.
4. Tanner Stage 1 breast development for females or Tanner Stage 1 external genitalia development for males at screening.
5. Ambulatory and able to stand without assistance.

Exclusion Criteria:

1. Bone age ≥14 years as assessed by the investigator based on hand and wrist X-ray taken within 6 months prior to Day 1.
2. Current evidence of growth plate closure (proximal tibia, distal femur), or AGV ≤ 1.5 cm/year over a period ≥6 months prior to screening.
3. Have a form of skeletal dysplasia other than ACH or known medical conditions that result in short stature or abnormal growth, including but not limited to severe achondroplasia with developmental delay and acanthosis nigricans (SADDAN), Turner syndrome, pseudoachondroplasia, inflammatory bowel disease, chronic renal insufficiency, active celiac disease a, Vitamin D deficiency b, untreated hypothyroidism c, poorly controlled diabetes (HbA1c ≥8.0%) or diabetic complications d.

   1. Celiac disease responsive to a gluten-free diet is allowed
   2. Vitamin D deficiency or insufficiency with a 25-hydroxyvitamin D [25- (OH) D] level ≥ 30 nmol/L after supplementation is allowed. Vitamin D deficiency is defined as 25-(OH) D level <30 nmol/L. Vitamin D insufficiency is defined as 25-(OH) D level 30~50 nmol/L. Patients with Vitamin D deficiency or insufficiency must be on Vitamin D regimen prior to screening
   3. Patients with hypothyroidism meeting the following criteria are allowed to enroll: must be clinically euthyroid for one month prior to screening and, in the opinion of the investigator, have achieved any catch-up growth expected from thyroxine replacement
   4. Patients with diabetes must have been on stable medication regimen for 3 months prior to screening
4. History or presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones.
5. Impaired cardiac function or clinically significant cardiovascular disease, including any one of the following: New York Heart Association class II or higher heart disease, congenital heart disease (patients with repaired uncomplicated patent ductus arteriosus or atrial/ventricular septal defect with repair are allowed), clinically significant arrhythmias requiring therapy, aortic regurgitation, congestive heart failure, or any other uncontrolled heart disease.
6. For ACH-related complications: Current severe sleep apnea, symptomatic and/or requiring intervention for hydrocephalus, or spinal cord compression at the cranio-cervical junction, and has previously undergone ventriculoperitoneal shunt surgery.
7. Bone fracture within 6 months prior to screening (within 2 months for finger and toe fractures).
8. Have received any dose of medications affecting stature or body proportionality, such as human growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids within 3 months prior to screening, or long-term treatment (>3 months) with the above drugs at any time.
9. Prior treatment with any CNP analogues or FGFR inhibitors. Prior use of any investigational drugs or investigational medical devices that affect stature or body proportionality.
10. Any comorbidities, disease or condition that, in the opinion of the investigator, may make the patient unlikely to fully complete the study-related procedures, may affect protocol compliance.

Ages: 30 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Achondroplasia
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2039-04-30 (Estimated)

PRIMARY OUTCOMES:
Annualized growth velocity (AGV) | Through the study completion, an average of three months, up to 2 years
  Annualized growth velocity (AGV)

SECONDARY OUTCOMES:
standing height | an average of three months, up to 2 years
  calculated to the nearest 0.1 cm
sitting height | an average of three months, up to 2 years
  calculated to the nearest 0.1 cm
sitting height to standing height ratio | an average of three months, up to 2 years
  This parameter is calculated as the ratio of sitting height to total standing height. It is used to assess the abnormality in body proportions, specifically the relative trunk-to-lower limb length. In patients with achondroplasia, this ratio is typically increased. Within the clinical trial, this measure is used to evaluate the treatment drug's effect on body proportions.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Lu, Study Director — 12B, Building 1, No 515, Huanke Road, Pudong New Area, Shanghai 201210, China
Locations (8):
- China (8):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Women and Childrens Medical Center, Guangzhou, Guangzhou
  - Henan Children's Hospital, Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xin Hua Hospital Affiliatod to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided